CLINICAL TRIAL: NCT00246623
Title: A Randomized, Open-Label, Multicenter Study Assessing the Effects of Forced Exubera Dose Titration on Glycemic Control in Patients With Suboptimally Controlled Type 2 Diabetes on Two or More Oral Antidiabetic Agents
Brief Title: US Inhaled Insulin Dose Titration Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171067
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exubera; Continuous Glucose Monitoring; Respiratory Physiological Phenomena; Nutrition Assessment

INTERVENTIONS:
Drug: Exubera (inhaled insulin)
Procedure: 8-point glucose diary (to assess pre- and post prandial glucoses)
Procedure: Meal Tolerance Test
Procedure: 24-hour continuous glucose monitoring (at select sites)
Procedure: Pulmonary Function Testing
Procedure: Hypoglycemic Event Monitoring
Procedure: Laboratory Assessments
Behavioral: Nutritional Counseling and Diabetes Education

SUMMARY:
This study will examine how to dose Exubera (inhaled insulin) in patients who are not well controlled on two or more diabetes pills. This study should show that a large number of patients enrolled in the study can reach the target Hemoglobin A1C levels (7% or less) that have been set by the American Diabetes Association (ADA). Target goals should be achieved by adjusting the Exubera dose either weekly or twice weekly. Patients will also receive nutritional counseling and diabetes education as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age >= 18 years and <= 80 years, with a diagnosis of type 2 diabetes made at least 6 months prior to study entry, with hemoglobin A1C 7.5-10%
* Currently treated with 2 or more oral antidiabetic agents (sulfonylureas, metformin, and/or thiazolidinediones)

Exclusion Criteria:

* Type 1 diabetes
* Smoking within the past 6 months or significant pulmonary diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with type 2 diabetes (A1C 7.5-10% on >= 2 oral agents) in each study arm (Exubera dosage adjusted 'once weekly' or 'twice weekly') that attain an A1C of <=7% with forced dose titration of Exubera at 6 months.

SECONDARY OUTCOMES:
Secondary endpoints include change in A1C, fasting and 2 hr PP glucose, 24-hr mean glucose measured by continuous glucose monitoring, weight, lipids, and markers of oxidative stress. Hypoglycemia will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Hayden, Idaho
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bennington, Vermont

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171067&StudyName=US+Inhaled+Insulin+Dose+Titration+Study